CLINICAL TRIAL: NCT06497023
Title: Multi-modality Radiomics Diagnostic Model Based on DCE-MRI and Ultrasound Images for Benign and Malignant Breast Lesion Classification
Brief Title: Radiomics Model Based on DCE-MRI and Ultrasound Images for Breast Lesion Classification
Status: Completed | Type: Observational
Sponsor: Ma Zhe (Other)
Responsible Party: Sponsor-Investigator, Ma Zhe, Director of Ultrasound, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2024(055)
Record Dates: First submitted 2024-06-23; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- maligant: female patients with maligant breast masses who underwent biopsy and/or surgical resection.
- benign: female patients with benign breast masses who underwent biopsy and/or surgical resection.

SUMMARY:
To develop and compare multi-modality radiomics models based on DCE-MRI, B-mode ultrasound (BMUS) and strain elastography (SE) images for classifying benign and malignant breast lesions.

DETAILED DESCRIPTION:
In this retrospective study,555 breast lesions from 555 patients who underwent DCE-MRI, BMUS and SE examinations were randomly divided into training (n =388) and testing (n = 167) datasets. Radiomics features were extracted from manually contoured images. The inter-class correlation coefficient (ICC), Mann-Whitney U test and the least absolute shrinkage and selection operator (LASSO) regression was applied for feature selection and radiomics signature building.Nine radiomics models including four single-modality radiomics models (DCE-3D, DCE-2D, BMUS, and SE), four multi-modality radiomics models (BMUS + SE, DCE-3D + BMUS, DCE-3D + SE, and DCE-3D+SE+BMUS), and the combination diagnostic model(clinical features and DCE-3D+SE+BMUS features) were developed and evaluated by their discrimination, calibration, and clinical usefulness.

ELIGIBILITY:
Inclusion Criteria:

Patients with breast lesions underwent biopsy or surgical resection between January 1, 2018 and March 30, 2024.

Exclusion Criteria:

1. pathologicalresult of biopsy or surgical specimen was unavailable for the target lesion;
2. patients without DCE-MRI, BMUS and SE examinations before biopsy or surgery within one month;
3. patients hadperformed radiotherapy, chemotherapy, or breast biopsy before MRI and ultrasound examinations;
4. patients without completeDICOM data for each examination;
5. patients with poor-qualityimages.

Ages: 15 Years to 80 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Patients with breast lesions attending the First Affiliated Hospital of Shandong First Medical University were selected
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of different diagnostic models | Immediately evaluated after the radiomcis diagnostic model was built
  The accuracy of nine diagnostic models, including four single-modality radiomics models (DCE-3D, DCE-2D, BMUS, and SE), four multi-modality radiomics models (BMUS + SE, DCE-3D + BMUS, DCE-3D + SE, and DCE-3D+SE+BMUS),and the combination diagnostic model is the ratio of the sum of True Positive and True Negative to the total of True Positive, True Negative, False Positive, and False Negative.

SECONDARY OUTCOMES:
Sensitivity of different diagnostic models | Immediately evaluated after the radiomcis diagnostic model was built
  The sensitivity of nine diagnostic models, four single-modality radiomics models (DCE-3D, DCE-2D, BMUS, and SE), including four multi-modality radiomics models (BMUS + SE, DCE-3D + BMUS, DCE-3D + SE, and DCE-3D+SE+BMUS), and the combination diagnostic model is the ratio of True Positive to the sum of True Positive and False Negative.

OTHER OUTCOMES:
Specificity of different diagnostic models | immediately evaluated after the combination diagnostic model was built
  The specificity of nine different diagnostic models, including four single-modality radiomics models (DCE-3D, DCE-2D, BMUS, and SE), four multi-modality radiomics models (BMUS + SE, DCE-3D + BMUS, DCE-3D + SE, and DCE-3D+SE+BMUS), and the combination diagnostic model is the ratio of True Negative to the sum of True Negative and False Positive.
PPV of different diagnostic models | immediately evaluated after the combination diagnostic model was built
  The PPV of nine different diagnostic models, including four single-modality radiomics models (DCE-3D, DCE-2D, BMUS, and SE), four multi-modality radiomics models (BMUS + SE, DCE-3D + BMUS, DCE-3D + SE, and DCE-3D+SE+BMUS),and the combination diagnostic model is the ratio of True Positive to the sum of True Positive and False Positive.
NPV of different diagnostic models | immediately evaluated after the combination diagnostic model was built
  The NPV of nine different diagnostic models, including four single-modality radiomics models (DCE-3D, DCE-2D, BMUS, and SE), four multi-modality radiomics models (BMUS + SE, DCE-3D + BMUS, DCE-3D + SE, and DCE-3D+SE+BMUS), and the combination diagnostic model is the ratio of True Negative to the sum of True Negative and False Negative.

CONTACTS AND LOCATIONS:
Locations (1):
- QianfoshanH, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Lack of resources or infrastructure: Sharing IPDs requires resources and infrastructure to ensure data security, manage access requests and provide necessary documentation. Currently these resources are not well developed, so it may be difficult to share IPDs.